CLINICAL TRIAL: NCT02287597
Title: An Observational Study of Avastin (Bevacizumab) in Patients With Metastatic Colorectal Cancer: Continued Avastin Plus Chemotherapy After First Progression in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29055
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This local, non-interventional, cohort study of patients with metastatic colorectal cancer (mCRC) will prospectively collect data from standard clinical practice of second-line treatment with chemotherapy plus Avastin (bevacizumab). There will be no additional diagnostic or therapeutic procedures required by this study, apart from those performed in everyday clinical practice for second-line treatment of mCRC in Croatia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >/=18 years
* Metastatic colorectal cancer (mCRC) previously treated with systemic treatment for advanced disease containing Avastin and chemotherapy; first-line Avastin received according to the Summary of Product Characteristics (SmPC)
* First line progression-free survival (PFS) >6 months
* Eligible for second-line chemotherapy regimen
* Period between first progression and start of second line treatment with Avastin and chemotherapy </=6 weeks

Exclusion Criteria:

* Contraindications, warnings and precautions for use specified in the Avastin SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer eligible for second-line chemotherapy and Avastin in Croatia.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Second-line time to progression, in months | Time between treatment initiation and tumor progression or death from cancer related cause, with censoring of patients who are lost to follow-up; up to 2 years

SECONDARY OUTCOMES:
Safety (composite outcome measure): Incidence of all adverse events, adverse events of special interest (AESI) for bevacizumab and pregnancies reported in second line mCRC treatment with Avastin plus chemotherapy | Up to 2 years
Safety (composite outcome measure): Incidence, nature and severity of all serious adverse events reported in second line mCRC treatment with Avastin plus chemotherapy and information on outcome and action taken with the drug | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Croatia (4):
  - Clinical Hospital Osijek; Dept For Oncology & Radiotherapy, Osijek
  - Uni Hospital Split; Oncology & Radiotherapy, Split
  - Clinical Hospital Centre Zagreb, Zagreb
  - Uni Hospital For Tumours; Dept of Medical Oncology, Zagreb